CLINICAL TRIAL: NCT01124032
Title: A Double Blind Crossover Study on the Effect of Methylphenidate on Decision-making Ability of Adults With ADHD Compared to Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Ziv Carmel,MD, shalvata Mental health center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHA 01-10
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADHD adults (Experimental)
  Interventions: Drug: methylphenidate
- healthy adults (Experimental)
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate — a capsule containing 20 mg

SUMMARY:
The study assesses the effect of Ritalin on working memory,attention,and decision-making measures in adults with ADHD and compares it to its effect on healthy adults, in a double-blind crossover design.We hypothesize that Ritalin will result in better performance in all measures,and that the improvement will be greater in the ADHD group.

ELIGIBILITY:
Inclusion Criteria:

* adults in the age of 21-50

Exclusion Criteria:

1. People diagnosed with a clinical disorder other than ADD/ADHD that may impair their performance in the tasks used in the study.
2. People for whom there is a contra-indication for consuming Ritalin.
3. Pregnant women and nursing women;

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
TOVA score | assessed twice, separated by 1-2 weeks.
IGT score | assessed twice, separated by 1-2 weeks
FPGT score | assessed twice, separated by 1-2 weeks
SWM score | assessed twice, separated by 1-2- weeks
digit span score | assessed twice, separated by 1-2- weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental Health center, Hod HaSharon, Israel

REFERENCES:
- [Background] Agay N, Yechiam E, Carmel Z, Levkovitz Y. Non-specific effects of methylphenidate (Ritalin) on cognitive ability and decision-making of ADHD and healthy adults. Psychopharmacology (Berl). 2010 Jul;210(4):511-9. doi: 10.1007/s00213-010-1853-4. Epub 2010 Apr 28. PMID 20424828